CLINICAL TRIAL: NCT03271541
Title: A Phase II, Single Arm, Multicenter, Proof-of-Mechanism Study to Investigate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of Bitopertin (RO4917838) in Adults With Non-Transfusion-Dependent Βeta-Thalassemia
Brief Title: A Study of Bitopertin (RO4917838) in Adults With Non-Transfusion-Dependent (NTD) Beta-Thalassemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP39642; 2016-004799-23 (EudraCT Number)
Record Dates: First submitted 2017-09-01; First posted 2017-09-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bitopertin (Experimental): Part 1 - The main study - 16 weeks in total:
  Participants will undergo a 6-week dose-escalation period followed by 10 weeks of treatment at the attained target dose of bitopertin.
  Part 2 - Open Label Extension (OLE) - up to an additional 12 months:
  Participants will be given the option to enroll into the OLE once the 16-week treatment of Part 1 has been completed.
  Participants who decide not to enroll in the OLE, at the end of Part 1 will enter a 6-week follow-up period.
  Interventions: Drug: Bitopertin

INTERVENTIONS:
Drug: Bitopertin — Bitopertin will be administered orally once daily at doses up to 120 milligrams (mg).
  Other Names: RO4917838

SUMMARY:
This proof-of-mechanism study is being performed to investigate the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of multiple oral doses of bitopertin in adults with NTD beta-thalassemia.

This study consists of two parts:

Part 1 - The main study - 16 weeks in total: Participants will undergo a 6-week dose-escalation period followed by 10 weeks of treatment at the attained target dose.

Part 2 - Open Label Extension (OLE) - up to an additional 12 months. Participants will be given the option to enroll into the OLE once the 16-week treatment of Part 1 has been completed. Participants who decide not to enroll in the OLE, at the end of Part 1 will enter a 6-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of beta-thalassemia
* Clinically defined non-transfusion-dependent anemia (Part 1 only), defined as Hb concentrations >7.5 grams per deciliter (g/dL) and <9.5 g/dL, less than or equal to 4 transfusions of red blood cell units within 1 year prior to study enrollment, and no transfusion within 12 weeks prior to study enrollment
* Completion of 16 weeks of treatment with bitopertin in Part 1 of this study with more than 80% compliance from expected use of study medication (based on patient diary and study drug accountability; Part 2 only)
* A favorable benefit-risk ratio from treatment with bitopertin as assessed by the Investigator (Part 2 only)

Exclusion Criteria:

* Any history of gene therapy
* History of hemolytic anemia except for beta-thalassemia
* Severe symptomatic splenomegaly and/or hepatomegaly with hypersplenism (Part 1 only)
* Any use of an erythropoiesis-stimulating agent within 24 weeks prior to enrollment.
* Initiation of iron chelation therapy or hydroxyurea within 24 weeks prior to enrollment (Part 1 only)
* Depression, treatment with anti-depressants, or other psychiatric illnesses and/or drug abuse
* Clinically significant/uncontrolled comorbid disease
* Pregnant or breastfeeding females
* Use of cytochrome P450 (CYP) 3A4 inhibitors within 2 weeks or CYP3A4 inducers within 4 weeks prior to study drug
* Active hepatitis B or C or known positive human immunodeficiency virus (HIV) test result
* Diagnosis of cancer within previous 5 years unless treatment has resulted in complete freedom from disease for at least 2 years
* Any major illness within 1 month or febrile illness within 1 week prior to study drug
* Pulmonary hypertension requiring oxygen therapy (Part 1 only)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Safety Outcome: Percentage of Participants with Adverse Events (AEs) - Part 1 only | Baseline, Week 16, up to Week 22
Efficacy Outcome: Change in Total Hemoglobin (Hb) Level from Baseline to End of 16-Week Treatment Period in Part 1 | Baseline to Week 16
Long-term Safety Outcome : Percentage of Participants with Adverse Events (AEs) - Part 2 only | Baseline to 19 Months

SECONDARY OUTCOMES:
Apparent Clearance of Bitopertin | Part 1: 2,12 hours (H) postdose (PD) on Day 1; 0 H predose (PRD) on Day 2; 0H PRD and 3H PD on Days 15,29,57; 0H PRD and 1,4H PD on Day 85; 0H PRD on Day 113; early withdrawal (ED) up to 22 wks. Part 2: 0H PRD and 1,4H PD on Days 183,365; ED up to 65 wks
Volume of Distribution of Bitopertin | Part 1: 2,12 hours (H) postdose (PD) on Day 1; 0 H predose (PRD) on Day 2; 0H PRD and 3H PD on Days 15,29,57; 0H PRD and 1,4H PD on Day 85; 0H PRD on Day 113; early withdrawal (ED) up to 22 wks. Part 2: 0H PRD and 1,4H PD on Days 183,365; ED up to 65 wks
Area Under the Concentration-Time Curve (AUC) of Bitopertin within a Dosing Interval | Part 1: 2,12 hours (H) postdose (PD) on Day 1; 0 H predose (PRD) on Day 2; 0H PRD and 3H PD on Days 15,29,57; 0H PRD and 1,4H PD on Day 85; 0H PRD on Day 113; early withdrawal (ED) up to 22 wks. Part 2: 0H PRD and 1,4H PD on Days 183,365; ED up to 65 wks
Minimum Observed Concentration (Cmin) of Bitopertin | Part 1: Predose (0 H) on Days 2, 15, 29, 57, 85, 113; and at early withdrawal (up to 22 weeks overall). Part 2: Predose (0 H) and postdose (1, 4 H) on Days 183, 365; and at early withdrawal (up to 65 weeks overall)
Maximum Observed Concentration (Cmax) of Bitopertin | Part 1: 2,12 hours (H) postdose (PD) on Day 1; 0 H predose (PRD) on Day 2; 0H PRD and 3H PD on Days 15,29,57; 0H PRD and 1,4H PD on Day 85; 0H PRD on Day 113; early withdrawal (ED) up to 22 wks. Part 2: 0H PRD and 1,4H PD on Days 183,365; ED up to 65 wks
Apparent Elimination Half-Life of Bitopertin | Part 1: 2,12 hours (H) postdose (PD) on Day 1; 0 H predose (PRD) on Day 2; 0H PRD and 3H PD on Days 15,29,57; 0H PRD and 1,4H PD on Day 85; 0H PRD on Day 113; early withdrawal (ED) up to 22 wks. Part 2: 0H PRD and 1,4H PD on Days 183,365; ED up to 65 wks
Accumulation Ratio of Bitopertin | Part 1: 2,12 hours (H) postdose (PD) on Day 1; 0 H predose (PRD) on Day 2; 0H PRD and 3H PD on Days 15,29,57; 0H PRD and 1,4H PD on Day 85; 0H PRD on Day 113; early withdrawal (ED) up to 22 wks. Part 2: 0H PRD and 1,4H PD on Days 183,365; ED up to 65 wks
Change from Baseline in Absolute Reticulocyte Count | Part 1: Baseline, Week 16. Part 2: Up to Week 65
Change from Baseline in Serum Lactate Dehydrogenase Level | Part 1: Baseline, Week 16. Part 2: Up to Week 65
Change from Baseline in Serum Bilirubin Level | Part 1: Baseline, Week 16. Part 2: Up to Week 65
Change from Baseline in Absolute Red Blood Cell Count | Part 1: Baseline, Week 16. Part 2: Up to Week 65
Change in Total Hb Level from Baseline to the End of the Treatment Period in Part 2 | Baseline, 19 Months

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (2):
  - Centro della Microcitemia e delle Anemie Congenite - Ospedale Galliera; Oncologia /Cardiologia, Genoa, Liguria
  - Ospedale Maggiore di Milano; Cardio-Metabolic Diseases, Milan, Lombardy
- Chronic Care Center, Baabda, Lebanon
- Siriraj Hospital; Division of Haematology-Oncology, Bangkok Noi, Thailand

REFERENCES:
- [Derived] Taher AT, Viprakasit V, Cappellini MD, Kraus D, Cech P, Volz D, Winter E, Nave S, Dukart J, Khwaja O, Koerner A, Hermosilla R, Brugnara C. Haematological effects of oral administration of bitopertin, a glycine transport inhibitor, in patients with non-transfusion-dependent beta-thalassaemia. Br J Haematol. 2021 Jul;194(2):474-477. doi: 10.1111/bjh.17479. Epub 2021 Apr 30. No abstract available. PMID 33931857